CLINICAL TRIAL: NCT00037687
Title: A Phase 3 Study to Demonstrate the Safety and Efficacy of Recombinant Platelet-Activating Factor Acetylhydrolase (rPAF-AH, Pafase®) for Reducing 28 Day All Cause Mortality in Patients With Severe Sepsis
Brief Title: Safety and Efficacy of Recombinant Human Platelet-Activating Factor Acetylhydrolase for the Treatment of Severe Sepsis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: ICOS Corporation (Industry)
Collaborators: Suntory Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAR03; BB-IND 9538
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-01

CONDITIONS: Sepsis
Keywords: Severe sepsis; Platelet-activating factor acetylhydrolase
MeSH Terms: conditions — Sepsis

INTERVENTIONS:
Drug: rPAF-AH

SUMMARY:
The objective of this study is to demonstrate that rPAF-AH is safe and reduces 28 day all cause mortality in patients with severe sepsis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter study of rPAF-AH compared to placebo in patients with severe sepsis. Eligible patients from investigative sites located throughout the United States and other countries will be randomized to receive either rPAF-AH or placebo administered daily for five consecutive days by intravenous (IV) infusion. All patients will be evaluated for safety and efficacy endpoints over 28 days. A follow-up evaluation will occur approximately 6 months after Day 28 to assess functional status and quality of life.

ELIGIBILITY:
Inclusion criteria

* Clinical diagnosis of severe sepsis
* At least 18 years old
* Patient or legally authorized representative able to provide informed consent

Exclusion criteria

* Severe lung injury (acute respiratory distress syndrome)
* Immunocompromised
* Severe liver disease
* Inflammation of the pancreas, organ rejection, or burns to more than 30% of body
* Enrolled in another clinical trial
* Already participated in this or other rPAF-AH study
* There is not a commitment to aggressive treatment
* Has a disease with life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500
Dates: Start 2001-04; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- Mary E. Lonien, M.S., Bothell, Washington, United States

REFERENCES:
- [Background] The Pafase Phase II ARDS Prevention Study Group. Recombinant platelet-activating factor acetylhydrolase (Pafase) decreases the incidence of acute respiriatory distress syndrome (ARDS) and 28 day all cause mortality (Abstract). Intensive Care Med (2000); 26: S321.